CLINICAL TRIAL: NCT00614510
Title: The SynCardia CardioWest Temporary Total Artificial Heart (TAH-t) Postmarket Surveillance Study
Brief Title: SynCardia CardioWest TAH-t Postmarket Surveillance Study
Status: Completed | Type: Observational
Sponsor: SynCardia Systems. LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: PR 05003; P030011/S1
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-03

CONDITIONS: Biventricular Failure

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CardioWest temporary Total Artificial Heart (TAH-t) — The SynCardia CardioWest temporary Total Artificial Heart (TAH-t) system is a pulsatile biventricular device that replaces a patient's native ventricles and valves and pumps blood to both the pulmonary and systemic circulation. The system consists of the implantable CardioWest TAH-t and an external console connected by drivelines.

SUMMARY:
The purpose of this study is to demonstrate that the results achieved in the original pivotal clinical investigation of 81 subjects from five clinical sites are generalizable to new clinical sites that complete the staff training defined in the SynCardia Systems, Inc. Training Manual and who enroll subjects who meet the intended use defined in the product Instructions for Use.

ELIGIBILITY:
Inclusion Criteria:

* The TAH-t is indicated for use as a bridge to transplant in cardiac transplant-eligible candidates at risk of imminent death from biventricular failure.

Exclusion Criteria:

* Patients who are not cardiac transplant eligible.
* Patients who do not have sufficient space in the chest area vacated by the natural ventricles. Generally this includes patients who have body surface areas <1.7m², or who have a distance between the sternum and the 10th anterior vertebral body measured by computed tomography imaging (CT scan) < 10 cm.
* Patients who cannot be adequately anticoagulated on the TAH-t.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been or will be implanted with the SynCardia Total Artificial Heart.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2006-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Subject survival at 30-days and one-year post transplant | 30-days and one-year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Jack G Copeland, MD, Principal Investigator — University Medical Center